CLINICAL TRIAL: NCT06212583
Title: A Randomized Trial of High-risK metachroNous oligometastatIc Prostate Cancer With hiGh-risk Mutations Treated witH meTastasiS Directed Therapy and Niraparib/Abiraterone Acetate and Prednisone (KNIGHTS)
Brief Title: High-Risk Metachronous Oligometastatic Prostate Cancer Trial
Acronym: KNIGHTS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Jason Molitoris, MD PhD, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00108148; GCC 23100 (Other: University of Maryland Medical System)
Record Dates: First submitted 2023-12-14; First posted 2024-01-19 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Oligometastatic Disease
MeSH Terms: conditions — Prostatic Neoplasms | interventions — niraparib; Abiraterone Acetate; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Androgen deprivation therapy + Stereotactic ablative radiation (Active Comparator)
  Interventions: Radiation: Stereotactic ablative radiation therapy (SABR); Drug: Androgen deprivation therapy (ADT)
- Androgen deprivation therapy + Stereotactic ablative radiation + niraparib/abiraterone acetate (Active Comparator)
  Interventions: Drug: niraparib/abiraterone acetate; Radiation: Stereotactic ablative radiation therapy (SABR); Drug: Androgen deprivation therapy (ADT)

INTERVENTIONS:
Drug: niraparib/abiraterone acetate — Patients on Arm 2 to receive drug for 6 months
  Arms: Androgen deprivation therapy + Stereotactic ablative radiation + niraparib/abiraterone acetate
Radiation: Stereotactic ablative radiation therapy (SABR) — Both arms will receive SABR
Drug: Androgen deprivation therapy (ADT) — All ADT is provided as best prescribed for patient per their medical oncologist.

SUMMARY:
The purpose of this research study is to compare the effects, good and/or bad, of using the standard of care treatment, hormonal therapy + Stereotactic Ablative Radiation (SABR) to the metastatic lesions, compared to standard of care and addition of 6-months of niraparib/abiraterone acetate combination pills and prednisone for participants with recurrent metastatic prostate cancer.

DETAILED DESCRIPTION:
In this trial all participants will be randomized to one of the two groups. You will be randomly assigned (by chance, like the flip of a coin) to one of the two groups: 1: Standard of care treatment (hormonal therapy + SABR to the metastatic lesions) or 2: Standard of care treatment + 6-months of niraparib/abiraterone acetate combination pills and prednisone. Participants in both groups will receive rectal swabs and various blood tests to assess circulating tumor cells, genomic sequencing, and tumor markers. Both groups will also participate in quality-of-life surveys

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age (or the local legal age of consent).
2. Patient must have at least one and up to three asymptomatic metastatic tumor(s) of the bone, soft tissue, or extra-pelvic nodal region each < 5 cm or < 250 cm3 that develop within the past 6-months that are seen on imaging. A nodal lesion is defined to include nodal conglomerates located in the same nodal chain such that they can be treated in one SABR field. Up to five lesions are allowed on advanced functional imaging such as fluciclovine (Axumin), choline or Prostate Specific Membrane Antigen (PSMA) PET-CT scan.

   1. CT or MRI scan within 6 months of enrollment
   2. Bone scan within 6 months of enrollment
   3. Fluciclovine (Axumin), choline, or PSMA PET-CT scan within 6 months of enrollment (PET-CT scan is reasonable for study entry imaging as an alternative to CT/MRI scan and bone scan)
3. Must have a high-risk pathogenic mutation (TP53, BRCA1/2, PALB2, ATM, BRIP1, CHEK2, FANCA, RAD51B, RAD54L, MUTYH) by next generation sequencing. ATM mutation enrollment will be capped at 5% of the overall population.
4. Histologic confirmation of prostate adenocarcinoma (primary or metastatic tumor).
5. Patient may have had prior systemic therapy and/or ADT so long as testosterone is > 100 ng/dl prior to enrollment
6. PSA > 0.5 but <50 at enrollment.
7. Prostate Specific Antigen Doubling Time (PSADT) < 15 months
8. Baseline testosterone > 100 ng/dl
9. Patient must have a life expectancy ≥ 12 months.
10. Patient must have an ECOG performance status ≤ 2.
11. Adequate hematologic, renal, and hepatic function at screening defined as follows:

    • Absolute neutrophil count ≥1.5 x 109/L

    • Hemoglobin ≥9.0 g/dL, independent of transfusions for at least 28 days
    * Platelet count ≥100 x 109/L
    * Creatinine <2 x upper limit of normal (ULN)
    * Serum potassium ≥3.5 mmol/L
    * Serum total bilirubin ≤1.5× ULN or direct bilirubin ≤1 x ULN (Note: In participants with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin, and if direct bilirubin is ≤1.5 × ULN, participant may be eligible)
    * AST or ALT ≤3 × ULN
12. Patient must have the ability to understand and the willingness to sign a written informed consent document
13. Able to swallow the study medication tablets whole.
14. While on study medication and for 4 months following the last dose of study medication, a male participant must agree to use condom and an adequate contraception method for female partner (WOCBP) A male participant must agree not to donate sperm while on study treatment and for a minimum of 4 months following the last dose of study medication.

<!-- -->

1. Castration-resistant prostate cancer (CRPC).
2. Prior radiation therapy to an overlapping site of a target lesion that would preclude further radiation therapy
3. Spinal cord compression or impending spinal cord compression.
4. Suspected intracranial and/or liver metastases (>10 mm in largest axis).
5. Patient receiving any other investigational agents.
6. Inability to receive any form of systemic therapy in the opinion of a treating medical oncologist.
7. Unable to lie flat during or tolerate PET/MRI, PET/CT or SABR.
8. Radiographical evidence of cranial parenchymal metastasis.
9. Active second primary malignancy; AML/MDS in medical history.
10. Uncontrolled hypertension and myocardial infarction/PE/cardiac failure in last 6 months.
11. Prior treatment with PARP inhibitor
12. Refusal to sign informed consent.
13. Pathological finding consistent with small cell or neuroendocrine carcinoma of the prostate.
14. History of adrenal dysfunction
15. Long-term use of systemically administered corticosteroids (>5mg of prednisone or the equivalent) during the study is not allowed. Short-term use (≤4 weeks, including taper) and locally administered steroids (eg, inhaled, topical, ophthalmic, and intra-articular) are allowed, if clinically indicated.
16. Active malignancies (ie, progressing or requiring treatment change in the last 24 months) other than the disease being treated under study. The only allowed exceptions are:

    * non-muscle invasive bladder cancer.
    * skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured.
    * malignancy that is considered cured with minimal risk of recurrence.
    * History or current diagnosis of MDS/AML.
17. Current evidence within 6 months prior to randomization of any of the following:

    • severe/unstable angina, myocardial infarction, symptomatic congestive heart failure,

    • clinically significant arterial or venous thromboembolic events (ie. Pulmonary embolism), or clinically significant ventricular arrhythmias.
18. Presence of sustained uncontrolled hypertension (systolic blood pressure >160 mm Hg or diastolic blood pressure >100 mm Hg). Participants with a history of hypertension are allowed, provided that blood pressure is controlled to within these limits by an antihypertensive treatment.
19. Known allergies, hypersensitivity, or intolerance to the excipients of niraparib/abiraterone acetate tablets
20. Current evidence of any medical condition that would make prednisone use contraindicated.
21. Received an investigational intervention (including investigational vaccines) or used an invasive investigational medical device within 30 days before the planned first dose of study medication.
22. Participants who have had the following ≤28 days prior to randomization:

    • A transfusion (platelets or red blood cells);

    • Hematopoietic growth factors;

    • Major surgery
23. Human immunodeficiency virus positive participants with 1 or more of the following:

    • Not receiving highly active antiretroviral therapy or on antiretroviral therapy for less than 4 weeks.
    * Receiving antiretroviral therapy that may interfere with the study medication
    * CD4 count <350 at screening.
    * An acquired immunodeficiency syndrome-defining opportunistic infection within 6 months of the start of screening.
    * Human immunodeficiency virus load >400 copies/mL
24. Active or symptomatic viral hepatitis or chronic liver disease; encephalopathy, ascites or bleeding disorders secondary to hepatic dysfunction.
25. Moderate or severe hepatic impairment (Class B and C per Child-Pugh classification system.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
PSA (Prostate Specific Antigen) evaluation at the 18-month progression of both treatment arms | 18 months
  PSA evaluation of progression at 18-month PSA , defined as PSA > 0.2 ng/mL in patients initially treated with radical prostatectomy and greater than nadir + 2 ng/mL for patients initially treated with definitive radiation, with testosterone >100 ng/dl of men who have oligometastatic castration-sensitive prostate cancer with high-risk mutations (TP53, BRCA1/2, PALB2, ATM, BRIP1, CHEK2, FANCA, RAD51B, RAD54L, MUTYH) treated with ADT + SABR MDT (6-mos) versus ADT + SABR MDT + niraparib/abiraterone acetate and prednisone (6-mos).

SECONDARY OUTCOMES:
Treatment-related adverse events of both treatment arms | 4 years
  Number of participants with treatment-related adverse events from ADT+ SABR MDT (6-mos) vs ADT + SABR MDT + niraparib/abiraterone acetate and prednisone (6-mos) in patients with metachronous oligometastatic CSPC disease.
Local control at 18 months after ADT+ SABR MDT (6-mos) vs ADT + SABR MDT + niraparib/abiraterone acetate and prednisone (6-mos) in patients with metachronous oligometastatic Castrate Specific Prostate Cancer (CSPC) disease. | 18 months
  Local control will be evaluated through clinical assessment and periodic imaging.
Time to locoregional progression, time to distant progression, time to new metastasis, radiographic progression-free survival and duration of response after randomization | 4 years
  Progression will be assessed for time to locoregional progression, time to distant progression, time to new metastasis, radiographic progression-free survival and duration of response after randomization.
Quality-of-life measured through EPIC tool following completion of ADT+ SABR MDT (6-mos) vs ADT + SABR MDT + niraparib/abiraterone acetate and prednisone (6-mos). | 4 years
  EPIC quality of life tool will be used to assess quality of life following treatment. Averages will be taken for each section in the survey (Urinary Function, Bowel Function, Sexual Function, and Hormonal function).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No